CLINICAL TRIAL: NCT06491875
Title: The Effect of Occupational Therapy and Sensory Integration Approach Supported Digital Storytelling on Facilitating Social Participation of Children With Autism Spectrum Disorder
Brief Title: The Effect of Digital Storytelling and Sensory Integration on Children With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Remziye Akarsu, Lecturer, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: akarsu
Record Dates: First submitted 2024-06-24; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism spectrum disorder; Sensory integration therapy; Digital storytelling
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autism Spectrum Disorder (Experimental): 1. Sensory integration training for children with ASD was conducted twice a week for two months (before Digital storytelling).
  2. The digital storytelling study was conducted for 16 hours over two months.
  Interventions: Behavioral: Digital Storytelling (DST); Behavioral: Sensory Integration Therapy (SIT)
- Typically Developing Children (Experimental): The digital storytelling study was conducted for 16 hours over two months.
  Interventions: Behavioral: Digital Storytelling (DST)

INTERVENTIONS:
Behavioral: Digital Storytelling (DST) — The DST activity emphasized the use of multimedia to bring the stories to life. At the beginning of the workshop, interactive circles were formed for informative interactions. Children with autism and typically developing children were asked to prepare a short video reflecting a personal experience from their own lives. The children's habits and interests were identified and they were made to work on preparing materials such as pictures, photographs, handicrafts, dough toys, etc. to be uploaded to the computer program. It was explained that they could also choose from ready-made photos in the video editing/editing program for their stories, and that they could make short audio recordings if they wished. Digital stories are usually prepared as videos that combine audio, video, and video clips to tell a story. The DST study was conducted for 16 hours over two months. During the DST, the mothers who wanted to participate and watch also participated in the study.
Behavioral: Sensory Integration Therapy (SIT) — Sensory integration training for children with ASD was conducted 2 days per week for 2 months. Taking into account the results of the Dunn Sensory Profile Scale, sensory approach strategies were determined for children with ASD, taking into account low and high neurological thresholds and hyper- and hyposensitive responses in the auditory, visual, tactile, vestibular and kinesthetic sensory systems. Sensory-motor activities with deep pressure and proprioceptive stimuli were used for children sensitive to tactile stimuli, and activities with linear and slow vestibular stimuli and resistive movement were used for children with kinesthetic sensitivity. In the intervention, swings, ball pools, ramps, rotation, and fast motion inputs were used in swing for children with hypersensitivity to motion, and sensory materials with different textures, play dough, and some other sensory materials were used for children with hypersensitivity to tactile sensory system.
  Arms: Autism Spectrum Disorder

SUMMARY:
Given the interest of children with Autism Spectrum Disorder (ASD) in using computers, this study examined the effect of Digital Storytelling (DST) activity on increasing activity participation and self-regulation. In this study, children with ASD and typically developing children were allowed to participate in DST workshops together. Selection of children intervention Children diagnosed with ASD and typically developing children attending Zeytinburnu Municipality Family Women Support and Disability Center (AKDEM) were included. The study was completed with a total of 15 children with ASD and 12 children with TD. In person-centered occupational therapy training with sensory integration, strategies including calming and reinforcing stimuli were identified to facilitate the social adaptation of children with autism and their participation in digital story activities. In the digital storytelling workshop, the Wevideo editing program was used. All participants were provided with an easy and fun application to express themselves by preparing stories with short videos about their lives, and the results were evaluated. This study emphasizes that children with autism spectrum disorder can successfully express their emotional expression skills and interests through digital stories. Digital stories are an essential tool to help these children express themselves. These findings may help educators and families working with children with ASD to develop new strategies to improve emotional expression skills and may serve as a basis for future studies.

DETAILED DESCRIPTION:
Introduction:

Occupational therapy is essential in addressing children's diverse needs and challenges to improve their overall health and quality of life. Occupational therapists working in pediatric settings focus on facilitating participation in meaningful activities in family, school, and community environments. To this end, occupational therapists play an essential role in ensuring that interventions are meaningful, engaging, and effective by selecting activities appropriate to children's individual needs and goals. These professionals work with children to improve their functional abilities in daily living tasks, education, and play, personalizing interventions to meet individual needs and promote independence. In this context, it can be said that occupational therapists realized the useful use of the digital storytelling technique in this study. Given the interest of children with Autism Spectrum Disorder (ASD) in using computers, this study examined the effect of Digital Storytelling (DST) activity on increasing activity participation and self-regulation.

Method Research design First, we made a selection of children diagnosed with ASD and typically developing children attending the Family Women Support and Disability Center (AKDEM) of Zeytinburnu Municipality. All registered families who had applied to the center for various reasons before and at the beginning of the research were informed about the research through face-to-face and telephone conversations, and they were all invited to participate. We then organized a training seminar to raise social awareness and inform the families of children with autism and typically developing children to participate.

The study consisted of three main data collections:

1. Assessment was conducted for 8 weeks, 5 days a week.
2. Sensory integration training for children with ASD was conducted 2 days a week for 2 months (before DST).
3. The DST study was conducted for 16 hours for 2 months.
4. The implementation results were conducted in 8 weeks, 5 days a week. AKDEM provided transportation for all children who volunteered for the study, and AKDEM health workers provided health care.

Setting As a preliminary study for the creation of the workshop, a suitable area in AKDEM was selected. Video creation programs to be used for DST were reviewed by the research team, and the We video program was selected for its ease of use and suitability for children with ASD. The research team s communication specialist provided training to the research team, educators, and professionals on the use of the We video program. Computers for use in the DST were provided by both institutions.

Study Participants The study included children with ASD and typically developing children of the same age. Children with ASD aged 7-11 years ( Mean 9,3) and typically developing children of similar age ( Mean 9,1) were included in the study. Inclusion criteria were that they came to AKDEM with a diagnosis of ASD according to DSM-5 criteria and that they were literate. Exclusion criteria were children reported by teachers at AKDEM to have maladaptive behaviors. At the beginning of the study, 16 children with ASD and 15 children with TD participated in the study, but later, 1 child from the ASD group and 3 children from the children with TD left the study. The study was completed with a total of 15 children with ASD and 12 children with TD, including 9 children with ASD and 7 children with TD at AKDEM and 6 children with ASD, and 5 children with TD at Biruni University SABIF Occupational Therapy Department.

Intervention Sensory integration education and strategies Sensory integration training for children with ASD was conducted 2 days per week for 2 months. Considering the Dunn Sensory Profile Scale results, sensory approach strategies were determined for children with ASD, taking into account low and high neurological thresholds and hyper- and hyposensitive responses in the auditory, visual, tactile, vestibular, and kinesthetic sensory systems. Sensory-motor activities with deep pressure and proprioceptive stimuli were used for children sensitive to tactile stimuli, and activities with linear and slow vestibular stimuli and resistive movement were used for children with kinesthetic sensitivity. In the intervention, swings, ball pools, ramps, rotation, and fast motion inputs were used in swing for children with hypersensitivity to motion, and sensory materials with different textures, play dough, and some other sensory materials were used for children with hypersensitivity to tactile sensory system.

In person-centered occupational therapy training with sensory integration, strategies including calming and reinforcing stimuli were determined to facilitate the social adaptation of children with autism and their participation in digital story activities. For children who are sensitive to visual and/or auditory stimuli, dimmer and quieter activity corners were planned for the DST study. Some children were placed on weight cushions on their knees during the DST. Strategies to facilitate their participation were identified, such as allowing them to jump on the trampoline when they wanted and allowing them to move to calm music or rhythm to facilitate their regulation. The intervention program was prepared and implemented by the Ayres SIPT-certified occupational therapists and physiotherapists in the research team, psychologists, counselor educators, and specialists working in the research team in consensus.

Considering the sensory integration and learning level of the child with autism, the materials to be used (play dough, handicraft, paper, cardboard, drawing pencils, paints, brushes, etc.) and guidance strategies (sound, light layout of the workshop, calming approach strategies) were determined for the digital storytelling application in cooperation with the occupational therapist, educator and communicator.

Digital Story Workshops In the digital storytelling workshops using the Wevideo editing program, all participants were provided with an easy and fun application to express themselves by preparing stories with short videos about their lives, and the results were evaluated. The research team's associate professor of communication trained the research team's trainers and counselors in the digital storytelling program. The study also trained children and their families to use the selected digital storytelling program. The DST activity emphasized the use of multimedia to bring the stories to life.

At the beginning of the workshop, interactive circles were formed for informative interactions. Children with autism and typically developing children were asked to prepare a short video reflecting a personal experience from their own lives. The children's interests were identified, and they were made to work on preparing materials such as pictures, photographs, handicrafts, dough toys, etc., to be uploaded to the computer program. It was explained that they could also choose from ready-made photos in the video editing/editing program for their stories and make short audio recordings if they wished. Digital stories are usually prepared as videos that combine audio, video, and video clips to tell a story. The DST study was conducted for 16 hours over two months. During the DST, the mothers who wanted to participate and watch participated in the study.

Data collection tools Measurement and evaluation methods realized in the research: Individual interviews with the families of children with autism, typically developing children (TD) were evaluated with the semi-structured interview method prepared by the research team. Data collection w s completed in 5 days with the semi-structured interview method about the perspectives of typically developing children and their families on autism and the difficulties they experience.

Assessing children with ASD Sensory characteristics of children with Autism Spectrum Diagnosis were evaluated with the Turkish version of the Dunn Sensory Profile created by Winne Dunn. Turkish adaptatio, reliability and validity were performed by Kayihan et al. Sensory Profile is a 125-question questionnaire filled out by parents used to measure the Sensory Processing characteristics of children aged 3-10 years. This questionnaire consists of 3 main sections and 14 different subsections. The first section Sensory Processing (6 subsections) measures children's response to a specific sensory input. The second section (Modulation (5 subsections) assesses children's ability to modulate sensory input in order to carry out activities of daily living. The third section (Behavioral and Emotional Reactions 3 subsections) assesses children's behavioral and emotional characteristics after processing sensory information. Each item of this test is scored between 1-5.

In our study, the Short Child Occupational Profile (SCOPE) is a scale that occupational therapists use. It defines the child's activity participation according to symptoms, diagnosis, and age. The child's skill, willpower, and habits are determined by their weaknesses and strengths. Environmental res, reactive, or facilitating aspects are examined. The SCOPE scale i a standardized measurement tool with Turkish validity and reliability that examines the child's participation in daily activities from a developmental perspective with 25 items in six sections. The first 5 sections (motivation, habit, communication) and interaction skills, process skills, and motor skills and their effects on participation performance are examined. The last section investigates how the environment affects the child's ability. Scoring is done through facilitators, allows, hinders, and restricts the child's participation in the activity. In our study, this scale was used to determine the personal and environmental factors related to children's activity participation.

In addition, the Child Occupational Self-Assessment Scale (COSA) was used. It is a Model of Human Occupation (MOHO) -base self-report scale used to measure children's perceived competence and the importance of their participation in daily activities. This assessment i suitable for children aged 6-17 years. The COSA consists of 25 items, and the child rates each statement using two 4-point Likert scales. For each item, one of the Likert scales measures the perceived level of efficacy for the reading with the statements: I have a lot of problems doing this, I have some problems doing this, I can do this well, and I can do this very well.

This study highlights that children with autism spectrum disorder can successfully express their emotional expression skills and interests through digital stories. Digital stories are seen as an important tool that can help these children express themselves. These findings may help educators and families working with children with ASD develop new strategies to improve emotional expression skills, and they may serve as a basis for future studies. Looking at the results of the scales administered at the end of the sensory integration intervention supported by DST, the results of the Dunn Sensory Profile Scale show that the sensory processing skills of children with ASD improved.

ELIGIBILITY:
Inclusion Criteria:

Getting diagnosed with ASD according to DSM-5 criteria

Knowing how to read and write

Exclusion Criteria:

Children reported by teachers to have maladaptive behavior

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-04-22 (Actual)

PRIMARY OUTCOMES:
The Short Child Occupational Profile | four weeks
  This scale is a tool that defines the child's occupational participation according to symptoms, diagnosis and age, and determines the child's skills, willpower and habits with their weaknesses and strengths. Environmental restrictive or facilitating aspects are examined. Scoring is made as follows: Facilitates the child's participation in the activity (4), Allows (3), Obstacles (2), Restrictions (1). As the scores increase, it is concluded that the occupational participation is good.
The Child Occupational Self Assessment Scale | four weeks
  It is a Model of Human Occupation (MOHO)-based self-report scale used to measure children's perceived competence and importance of their participation in daily activities. This assessment is suitable for children aged 6-17 years. The COSA consists of 25 items and the child rates each statement using two 4-point Likert scales. Higher scores indicate better occupational performance.

SECONDARY OUTCOMES:
The Sensory Profile | four weeks
  Sensory Profile is a measurement tool used to evaluate sensory modulation. A 125-question questionnaire filled out by parents was used to measure the sensory processing characteristics of children aged 3-10 years. This questionnaire consists of 3 main sections and 14 different subsections. 3 main sections are, Sensory Processing, Modulation and Behavioral and Emotional Responses. Each item of this test is scored between 1-5.and 14 different subsections. The first section Sensory Processing (6 subsections) measures children's response to a specific sensory input. The second section (Modulation (5 subsections) assesses children's ability to modulate sensory input in order to carry out activities of daily living. The third section (Behavioral and Emotional Reactions 3 subsections) assesses children's behavioral and emotional characteristics after processing sensory information. Each item of this test is scored between 1-5.Higher scores indicate better sensory processing.

CONTACTS AND LOCATIONS:
Locations (1):
- Remziye Akarsu, Istanbul, Turkey (Türkiye)